CLINICAL TRIAL: NCT04469881
Title: Netflix Streaming Services in the Operating Room During Total Knee Replacement - a Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost research staff - unable to enroll until new research staff is hired.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20017126
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (Experimental): Wear VR glasses and watch movies during surgery
  Interventions: Behavioral: VR

INTERVENTIONS:
Behavioral: VR — Participants will be asked to do the following things:
  1. Wear VR goggles for the duration of the surgery
  2. Answer questions about their experience with the VR goggles
  3. Give permission for the researchers to collect information about the anesthesia medications used, pain medications used, and reported pain scores during the surgery and during recovery in the hospital

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of watching streamed videos through virtual reality (VR) goggles during surgery.

The results of this study will be used to evaluate whether video-streaming services on VR goggles are worthwhile additions to standard anesthesia care during total knee surgery.

DETAILED DESCRIPTION:
Usual anesthetic care for total knee replacement involves intravenous sedation as well as spinal anesthesia. In this study, participants will receive usual care, and in addition, will be asked to wear VR goggles once they arrive in the operating room. Participants will choose from a selection of 10 shows and movies to watch for the duration of the surgery (approximately 2 hours).

ELIGIBILITY:
Inclusion Criteria:

1. undergoing a primary elective total knee replacement by one of the orthopedic joint surgeons at Virginia Commonwealth University Medical Center
2. 18 years of age or older
3. eligible for spinal anesthesia
4. mentally capable of understanding instructions on how to request anesthesia medication

Exclusion Criteria:

1. identified as a member of regulated vulnerable population
2. ineligibility for spinal anesthesia
3. morbid obesity (body mass index greater than 40)
4. allergy to propofol or midazolam
5. pre-operative daily opioid consumption of more than 10 mg oxycodone every 6 hours (over 60 morphine miligram equivalents per day)
6. daily benzodiazepine consumption
7. history of alcohol or recreational drug abuse
8. hearing or visually impaired individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Sedation requirement | approximately 2 hours
  Micrograms of propofol per kilogram per minute

SECONDARY OUTCOMES:
Participant pain rating | 24 hours
  Average pain score measured immediately after surgery and every 4 hours afterwards for 24 hour. Pain will be rated on a 0 to 10 scale with 0 being no pain and 10 being the worst pain imaginable.
Opioid consumption | 24 hours
  Total miligram morphine equivalents of opioid pain medication administered during 24 hours post surgery.
Time to first opioid request | up to 24 hours
  Time in minutes between leaving the operating room and administration of first oral opioid.

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Tran, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No